CLINICAL TRIAL: NCT00615771
Title: Embryo Transfer on Day 2 vs. Day 3 After Oocyte Retrieval in Patients Who Plan to Replace All Embryos After an In Vitro Fertilization Cycle
Brief Title: Day of Embryo Transfer for Patients Undergoing In Vitro Fertilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Ruth Bunker Lathi, associate professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-01312008-991
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2011-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Day 2 embryo transfer (Experimental): Embryos are transferred 2 days after fertilization.
  Interventions: Procedure: Day 2 embryo transfer
- Day 3 embryo transfer (Active Comparator): Standard of care for women undergoing IVF with a limited number of embryos is to transfer all embryos on Day 3 after fertilization
  Interventions: Procedure: Day 3 embryo transfer

INTERVENTIONS:
Procedure: Day 3 embryo transfer — Standard of care
  Arms: Day 3 embryo transfer
Procedure: Day 2 embryo transfer — Embryos are transferred 1 day prior to standard of care
  Arms: Day 2 embryo transfer

SUMMARY:
We are examining whether pregnancy rates differ based on day of embryo transfer in patients who replace all available embryos after an In vitro Fertilization (IVF) cycle. Patients must be undergoing IVF treatment at Stanford University and patients will not receive compensation for their participation (no medical costs covered or patient payment for participation).

DETAILED DESCRIPTION:
The decision on the number of embryos to transfer after an IVF cycle is based on the number of available embryos, the quality of the embryos, the patient's age, and the goal of limiting multiple gestations. Stanford Fertility Center and most IVF centers examine the embryos on the third day after oocyte (egg) retrieval to select for the best quality embryos to transfer, and depending on quality, the remaining embryos are frozen to be used in the future. Patients with a limited number of embryos, those that plan to replace all available embryos after an IVF cycle, do not need to wait until the third day after oocyte retrieval to select embryos, and may replace the embryos on the second day after the oocyte retrieval. We are examining whether pregnancy rates differ among these patients based on the day of embryo transfer (Day 2 vs. Day3). Patients must be undergoing IVF treatment at Stanford University and patients will not receive compensation for their participation (no medical costs covered or patient payment for participation).

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing fresh IVF cycle at Stanford Fertility Center who plan on replacing all available embryos.

Exclusion Criteria:

Patients that do not meet above criteria.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 242 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pregnancy rates | 1 year

SECONDARY OUTCOMES:
Live birth rates | 1 year
Multiple gestation rates | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lora K Shahine, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States